CLINICAL TRIAL: NCT02596334
Title: Randomized Clinical Trial to Evaluate the Efficacy of a Dolutegravir Monotherapy (Tivicay®) Versus the Maintenance of a Successful Triple Therapy Using Abacavir + Lamivudine + Dolutegravir (Triumeq®) in HIV-1- Infected Patients
Brief Title: Study to Evaluate the Efficacy of MONotherapy of TiviCAY® Versus a Triple Therapy in HIV-1-infected Patients
Acronym: MONCAY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: 5 patients on tivicay had virological failure
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRO 2015-03
Record Dates: First submitted 2015-10-16; First posted 2015-11-04 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: HIV
Keywords: HIV-1 infected patient; monotherapy; dolutegravir
MeSH Terms: interventions — dolutegravir; abacavir; Lamivudine; abacavir, dolutegravir, and lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- triple therapy (Active Comparator): dolutegravir + abacavir + lamivudine (TRIUMEQ) : oral administration, one tablet daily during 48 weeks.
  Interventions: Drug: dolutegravir 50mg +abacavir 600mg +lamivudine 300mg
- monotherapy (Experimental): dolutegravir (TIVICAY) : 50 mg, oral administration, one tablet daily during 48 weeks.
  Interventions: Drug: dolutegravir

INTERVENTIONS:
Drug: dolutegravir 50mg +abacavir 600mg +lamivudine 300mg
  Other Names: Triumeq, EU/1/14/940/001
  Arms: triple therapy
Drug: dolutegravir
  Other Names: Tivicay , EU/1/13/892/001
  Arms: monotherapy

SUMMARY:
Triple antiretroviral regimens have greatly improved the prognosis of patients living with HIV (PLHIV). Patients virologically controlled and having a good immune restoration can have a life expectancy close or equal to that of people not infected with HIV.[1] However, this is under the condition of a "lifetime" maintenance of an undetectable plasma viral load (pVL) (<50 cp/ml). On the other hand it is well established that aging increases comorbidities among PLHIV and the burden of co-medications.[2] This also has the consequence of frequent drug-drug interactions. In this context it is important to decrease pills burden, side-effects and drug-drug interactions, while maintaining undetectability.

Currently, there is a strong interest for medical research to validate lightened regimens (i.e. bithérapies [3-7] and monothérapies [8,9], particularly in a maintenance strategy, with the primary objective of reducing burden of pills and side effects. Several monotherapy trials using a boosted protease inhibitor (PI/r) showed high level of viral suppression, even if this proportion was not always non-inferior to maintaining a triple therapy. [8,9] Fortunately, when virological failure occurred under monotherapy virologic suppression was easily restored by the addition of two NRTI. Patients who are most likely to maintain viral suppression under a reduced scheme are those that have a high nadir (> 100 CD4 / mm3), no previous AIDS event and a sustained virologic suppression (>12 months).

Monotherapy is the option that best reduces the burden of pills and the risk of side effects or drug-drug interactions. It must be considered using very powerful molecule that harbor a strong binding to its ligand in order to minimize the risk of selecting resistant mutants in the case of virologic failure. To be as simple as possible in its use, it must be a single agent administered as a single dose once a day and not boosted if possible. The molecule must have very good tolerance. Finally, to be effective in viral sanctuaries this molecule should have a good (or sufficient) diffusion to ensure effective Cmin on wild viral strains. Dolutegravir meets all these exigences.[10] In addition, our team recently presented results of a pilot study showing that the switch of a successful combined antiretroviral regimen to dolutegravir monotherapy maintained undetectable viral load (<20 cp/ml) after a median of 7 months (range 6.5-10 months).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1-infected patients with no previous AIDS event (excluding a healed tuberculosis);
* Current antiretroviral treatment associating dolutegravir + abacavir + lamivudine for at least 1 month;
* Nadir CD4 ≥ 100/mm3;
* Plasma RNA viral load < 50 copies/ml for at least 12 months;
* Plasma RNA viral load <20 or 40 copies/ml (according to the threshold of the method used by local laboratory) at the screening visit;
* No documented virologic failure or known resistance to any integrase inhibitor,
* Patient having provided a written consent;
* Patients follow-up possible in ambulatory;
* Patient age > 18 years;
* Covered by health insurance

Exclusion Criteria:

* Non-compliant patient

  * Subject is pregnant, or lactating, or of childbearing potential and without contraception;
  * Active opportunistic infections (defining AIDS);
  * Known hypersensibility to abacavir or lamivudine or dolutegravir;
  * Patients harboring HLA B*5701;
  * Major overweight (BMI ≥ 40);
  * Weight <40 kg;
  * Creatinine clearance < 50ml/min;
  * Cirrhosis or severe liver failure (factor V < 50%);
  * Life Prognosis threatened within 6 months;
  * Circumstances that may impair judgment or understanding of the information given to the patient;
  * Co-medication with carbamazepin, oxcarbamazepin, fosphenytoïn, phenobarbital, phenytoïn, primidon, St John's wort or dofetilid;
  * Malabsorption syndromes;
  * The following laboratory criteria:

    * Serum AST,ALT > 5 x upper limit of normal (ULN)
    * Thrombocytopenia with platelet count < 50.000/ml
    * Anemia with hemoglobin < 8g/dl
    * Polynuclear neutrophil count < 500/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2018-06-23 (Actual)

PRIMARY OUTCOMES:
Viral Load | Week 24
  Percentage of patients having a viral load <50 copies/ml in each arm at week 24

SECONDARY OUTCOMES:
Viral load | between Week 4 and Week 48
  Percentage of patients having a confirmed viral load > 50 copies/ml between week 4 and week 48
Delta CD 4 | until Week 48
  delta CD4 in each arms from Baseline to W48, comparison between arms
Residual activation measures (sub study) | Week 24
  CD4+CD38+DR+, CD8+CD38+DR+
Residual activation marker measures (sub study) | Week 24
  sCD14, sCD163,
Pro-inflammatory cytokins measures (sub study) | Week 24
  TNFα, IFNγ, IL6, IP-10
Inflammatory marker measures (sub study) | Week 24
  CRPus
virus genotype | Until Week 48
  Evolution of viruses genotype profiles of patients who present a virologic failure
RNA and DNA viral load (sub study) | Week 24 to week 48
  RNA and DNA viral load in the genital tract (cervico-vaginal secretions or sperm): comparison between arms
HIV DNA evolution | between day 0 and week 48
  HIV DNA evolution in each arm from baseline to W48; comparison between arms
Virological failure predictive factors | 48 weeks
  Determination of virological failure predictive factors
Impact of the strategy on the acceptability and quality of life | 48 weeks
  determination of quality of life with questionnary, comparison between arms
Proportion of patients with an adverse event | 48 weeks
Proportion of patients with a severe adverse event | 48 weeks
Creatinine clearance change | 48 weeks
  Biological parameters evolution in each arm
Lipidic profiles | 48 weeks
  Biological parameters evolution in each arm
Clinical events | 48 weeks
  Clinical events with progression to AIDS or death. Proportion of individuals developing a new CDC-event (as defined by cdc 1993 classification) from baseline to week 48.

CONTACTS AND LOCATIONS:
Overall Officials: HOCQUELOUX Laurent, Study Director — CHR d'ORLEANS
Locations (9):
- France (9):
  - CHD de VENDEE, La Roche-sur-Yon
  - CH de LA ROCHELLE, La Rochelle
  - CHRU de NANTES, Nantes
  - CH de NIORT, Niort
  - CHR d'ORLEANS, Orléans
  - CHRU de POITIERS, Poitiers
  - CHU de STRASBOURG, Strasbourg
  - CHRU de TOURS, Tours
  - CHU de NANCY, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] May MT, Gompels M, Delpech V, Porter K, Orkin C, Kegg S, Hay P, Johnson M, Palfreeman A, Gilson R, Chadwick D, Martin F, Hill T, Walsh J, Post F, Fisher M, Ainsworth J, Jose S, Leen C, Nelson M, Anderson J, Sabin C; UK Collaborative HIV Cohort (UK CHIC) Study. Impact on life expectancy of HIV-1 positive individuals of CD4+ cell count and viral load response to antiretroviral therapy. AIDS. 2014 May 15;28(8):1193-202. doi: 10.1097/QAD.0000000000000243. PMID 24556869
- [Background] Nachega JB, Parienti JJ, Uthman OA, Gross R, Dowdy DW, Sax PE, Gallant JE, Mugavero MJ, Mills EJ, Giordano TP. Lower pill burden and once-daily antiretroviral treatment regimens for HIV infection: A meta-analysis of randomized controlled trials. Clin Infect Dis. 2014 May;58(9):1297-307. doi: 10.1093/cid/ciu046. Epub 2014 Jan 22. PMID 24457345
- [Background] Cahn P, Andrade-Villanueva J, Arribas JR, Gatell JM, Lama JR, Norton M, Patterson P, Sierra Madero J, Sued O, Figueroa MI, Rolon MJ; GARDEL Study Group. Dual therapy with lopinavir and ritonavir plus lamivudine versus triple therapy with lopinavir and ritonavir plus two nucleoside reverse transcriptase inhibitors in antiretroviral-therapy-naive adults with HIV-1 infection: 48 week results of the randomised, open label, non-inferiority GARDEL trial. Lancet Infect Dis. 2014 Jul;14(7):572-80. doi: 10.1016/S1473-3099(14)70736-4. Epub 2014 Apr 27. PMID 24783988
- [Background] Prazuck T, Zucman D, Avettand-Fenoel V, Ducasse E, Bornarel D, Mille C, Rouzioux C, Hocqueloux L. Long-term HIV-1 virologic control in patients on a dual NRTI regimen. HIV Clin Trials. 2013 May-Jun;14(3):120-6. doi: 10.1310/hct1403-120. PMID 23835514
- [Background] Reynes J, Lawal A, Pulido F, Soto-Malave R, Gathe J, Tian M, Fredrick LM, Podsadecki TJ, Nilius AM. Examination of noninferiority, safety, and tolerability of lopinavir/ritonavir and raltegravir compared with lopinavir/ritonavir and tenofovir/ emtricitabine in antiretroviral-naive subjects: the progress study, 48-week results. HIV Clin Trials. 2011 Sep-Oct;12(5):255-67. doi: 10.1310/hct1205-255. PMID 22180523
- [Background] Calin R, Paris L, Simon A, Peytavin G, Wirden M, Schneider L, Valantin MA, Tubiana R, Agher R, Katlama C. Dual raltegravir/etravirine combination in virologically suppressed HIV-1-infected patients on antiretroviral therapy. Antivir Ther. 2012;17(8):1601-4. doi: 10.3851/IMP2344. Epub 2012 Sep 3. PMID 22941896
- [Background] Monteiro P, Perez I, Laguno M, Martinez-Rebollar M, Gonzalez-Cordon A, Lonca M, Mallolas J, Blanco JL, Gatell JM, Martinez E. Dual therapy with etravirine plus raltegravir for virologically suppressed HIV-infected patients: a pilot study. J Antimicrob Chemother. 2014 Mar;69(3):742-8. doi: 10.1093/jac/dkt406. Epub 2013 Oct 14. PMID 24128667
- [Background] Katlama C, Valantin MA, Algarte-Genin M, Duvivier C, Lambert-Niclot S, Girard PM, Molina JM, Hoen B, Pakianather S, Peytavin G, Marcelin AG, Flandre P. Efficacy of darunavir/ritonavir maintenance monotherapy in patients with HIV-1 viral suppression: a randomized open-label, noninferiority trial, MONOI-ANRS 136. AIDS. 2010 Sep 24;24(15):2365-74. doi: 10.1097/QAD.0b013e32833dec20. PMID 20802297
- [Background] Arribas JR, Horban A, Gerstoft J, Fatkenheuer G, Nelson M, Clumeck N, Pulido F, Hill A, van Delft Y, Stark T, Moecklinghoff C. The MONET trial: darunavir/ritonavir with or without nucleoside analogues, for patients with HIV RNA below 50 copies/ml. AIDS. 2010 Jan 16;24(2):223-30. doi: 10.1097/QAD.0b013e3283348944. PMID 20010070
- [Background] Greig SL, Deeks ED. Abacavir/dolutegravir/lamivudine single-tablet regimen: a review of its use in HIV-1 infection. Drugs. 2015 Apr;75(5):503-14. doi: 10.1007/s40265-015-0361-6. PMID 25698454
- [Derived] Hocqueloux L, Gubavu C, Prazuck T, De Dieuleveult B, Guinard J, Seve A, Mille C, Gardiennet E, Lopez P, Rouzioux C, Lefeuvre S, Avettand-Fenoel V. Genital Human Immunodeficiency Virus-1 RNA and DNA Shedding in Virologically Suppressed Individuals Switching From Triple- to Dual- or Monotherapy: Pooled Results From 2 Randomized, Controlled Trials. Clin Infect Dis. 2020 Apr 15;70(9):1973-1979. doi: 10.1093/cid/ciz511. PMID 31350995
- [Derived] Hocqueloux L, Raffi F, Prazuck T, Bernard L, Sunder S, Esnault JL, Rey D, Le Moal G, Roncato-Saberan M, Andre M, Billaud E, Valery A, Avettand-Fenoel V, Parienti JJ, Allavena C; MONCAY study group. Dolutegravir Monotherapy Versus Dolutegravir/Abacavir/Lamivudine for Virologically Suppressed People Living With Chronic Human Immunodeficiency Virus Infection: The Randomized Noninferiority MONotherapy of TiviCAY Trial. Clin Infect Dis. 2019 Oct 15;69(9):1498-1505. doi: 10.1093/cid/ciy1132. PMID 30601976